CLINICAL TRIAL: NCT02536287
Title: Comparison of Total Parathyroidectomy With Autotransplantation Versus Total Parathyroidectomy Without Autotransplantation:A Randomized Clinical Trial
Brief Title: Comparison of Total Parathyroidectomy With and Without Autotransplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, xpgeng, vice-president, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ahykdxdefsyy12
Record Dates: First submitted 2015-08-22; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Secondary Hyperparathyroidism
Keywords: secondary hyperparathyroidism; total parathyroidectomy; autotransplantation; morbidity; recurrence; postoperative hypocalcemia
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Recurrence | interventions — Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- total PTX without autotransplantation (Experimental): all parathyroid glands were found and removed
  Interventions: Procedure: total PTX without autotransplantation
- total PTX with autotransplantation (Active Comparator): all parathyroid glands were found and removed,and then a portion of it is sliced into 1*1*1 mm pieces for autotransplantation
  Interventions: Procedure: total PTX with autotransplantation

INTERVENTIONS:
Procedure: total PTX without autotransplantation — All parathyroid glands were found and removed and sent for histological confirmation,but without autotransplantation.
  Arms: total PTX without autotransplantation
Procedure: total PTX with autotransplantation — All parathyroid glands were found and removed and sent for histological confirmation,and then a portion of the smallest, preferably nonnodular parathyroid gland was chosen for autotransplantation,sliced into pieces measuring 1*1 *1 mm,and placed into the subcutaneous of the forearm.
  Arms: total PTX with autotransplantation

SUMMARY:
The purpose of this study is to compare short-term and long-term efficacy of total parathyroidectomy with autotransplantation and total parathyroidectomy without autotransplantation for Secondary hyperparathyroidism.

DETAILED DESCRIPTION:
Background:Secondary hyperparathyroidism (SHPT) is a common disorder in patients with chronic kidney disease. It is caused by permanent stimulation of the orthotopic and heterotopic parathyroid tissue due to phosphate retention, hypocalcemia, and vitamin D insufficiency. Despite the initiation of new therapeutic agents, several patients will require parathyroidectomy.There are three options for the surgical treatment of SHPT:subtotal PTX (3.5-gland resection,SPTX), total PTX with autotransplantation(TPTX+AT), and total PTX without autotransplantation(TPTX).SPTX and TPTX+AT both leave a fragment of activated,proliferated parathyroid tissue.Since the pathophysiological condition of chronic renal failure and maintenance dialysis continues, the growth stimulus persists and may cause recurrent sHPT.The SPTX procedure has a lesser likelihood of a non-functioning remnant, but recurrent disease always requires a neck reoperation that carries a high likelihood of recurrent laryngeal nerve palsy.Therefore most surgeons believe that TPTX+AT is a better procedure for patients with SHPT.

Because of the potential complication of permanent hypocalcemia and adynamic bone disease,TPTX was not introduced into clinical practice.However,recent retrospective studies demonstrated patients after TPTX did not develop permanent hypoparathyroidism and adynamic bone disease as initially expected.Postoperative hypocalcemia is temporary.TPTX may provide an alternative strategy to the currently performed procedures mainly because of the reported lower recurrence rates.An 8-year follow-up study showed the recurrence rates after TPTX is 7%.Recurrence rates after TPTX+AT is 21.4%,and the site of recurrence is located in approximately 80% at the graft and in 20% in the neck.However, to the present there is no randomized controlled trial to Compare the effects of total parathyroidectomy with autotransplantation and total parathyroidectomy without autotransplantation.The purpose of this study is to evaluate the short-term and long-term efficacy of total parathyroidectomy without autotransplantation comparison to total parathyroidectomy with autotransplantation.

Intervention: One hundred patients with SHPT need undergo parathyroidectomy at the Second Hospital of Anhui medical university were selected and divided into total parathyroidectomy without autotransplantation group and total parathyroidectomy with autotransplantation group, each group contains 50 cases.

Results:

1. Clinical data include: intact parathyroid hormone,serum calcium,serum phosphorus,calcium-phosphorus product,hemoglobin,operation time,morbidity,mortality,clinical symptoms and signs,recurrence and reoperation,quality of life scores.
2. Statistical method: groups t-test, analysis of variance were used.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female, aged 18 or older;
* Intact parathyroid hormone(iPTH) is more than 9 times the upper limit of the normal range (about 600pg/ml), with hypercalcemia or hyperphosphatemia;
* Refractory to medical therapy;
* Provided written informed consent.

Exclusion Criteria:

* Primary or tertiary hyperparathyroidism;
* Familial hyperparathyroidism (MENⅠ, MENⅡ, hereditary HPT);
* Neck surgical exploration history;
* Parathyroid malignant tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of intact parathyroid hormone(iPTH) | 1 day,1 week,1,3,6,12,18 and 24months
  Intact parathyroid hormone was collected before operation,1 day,1 week,1 month,3 months,6 months,12 months,18 months and 24months after the operation

SECONDARY OUTCOMES:
Change of serum calcium | 1 day,1 week,1,3,6,12,18 and 24months
  Serum calcium was collected before operation,1 day,1 week,1 month,3 months,6 months,12 months,18 months and 24months after the operation
Change of serum phosphorus | 1 day,1 week,1,3,6,12,18 and 24months
  Serum phosphorus was collected before operation,1 day,1 week,1 month,3 months,6 months,12 months,18 months and 24months after the operation
Change of calcium-phosphorus product | 1 day,1 week,1,3,6,12,18 and 24months
  Serum calcium*serum phosphorus was collected before operation,1 day,1 week,1 month,3 months,6 months,12 months,18 months and 24months after the operation
Change of hemoglobin | 1 day,1 week,1,3,6,12,18 and 24months
  Hemoglobin was collected before operation,1 day,1 week,1 month,3 months,6 months,12 months,18 months and 24months after the operation
Operation time | an expected average of 1.5 hours
  Operation time is defined as from skin incision to placement of last skin staple
Morbidity | 30 days
  The severity of complications was graded according to the Clavien-Dindo classification,The most common complication was recurrent laryngeal nerve palsy
Mortality | 30 days
  Operative mortality was defined as any death resulting from a complication during surgery
Clinical symptoms and signs | From 1 day after the operation, assessed up to 2 years
  Postoperative symptom relief was investigated
Recurrence and reoperation | From 1 day after the operation, assessed up to 2 years
  Recurrence and reoperation were recorded
Change of quality of life | 1year,2 years
  The Kidney Disease Quality of Life Short Form(KDQOL-SFTM) scale was used to evaluate quality of life before operation, 1 year and 2 years after parathyroidectomy

CONTACTS AND LOCATIONS:
Overall Officials: xiaoping geng, professor, Principal Investigator — the vice President of the second affiliated hospitalof Anhui medical university
Locations (1):
- the Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Result] Puccini M, Carpi A, Cupisti A, Caprioli R, Iacconi P, Barsotti M, Buccianti P, Mechanick J, Nicolini A, Miccoli P. Total parathyroidectomy without autotransplantation for the treatment of secondary hyperparathyroidism associated with chronic kidney disease: clinical and laboratory long-term follow-up. Biomed Pharmacother. 2010 May;64(5):359-62. doi: 10.1016/j.biopha.2009.06.006. Epub 2009 Oct 23. PMID 20435429
- [Result] Jia X, Wang R, Zhang C, Cui M, Xu D. Long-Term Outcomes of Total Parathyroidectomy With or Without Autoimplantation for Hyperparathyroidism in Chronic Kidney Disease: A Meta-Analysis. Ther Apher Dial. 2015 Oct;19(5):477-85. doi: 10.1111/1744-9987.12310. Epub 2015 May 6. PMID 25950238
- [Result] Tominaga Y, Matsuoka S, Sato T. Surgical indications and procedures of parathyroidectomy in patients with chronic kidney disease. Ther Apher Dial. 2005 Feb;9(1):44-7. doi: 10.1111/j.1774-9987.2005.00213.x. PMID 15828905
- [Result] Tominaga Y, Uchida K, Haba T, Katayama A, Sato T, Hibi Y, Numano M, Tanaka Y, Inagaki H, Watanabe I, Hachisuka T, Takagi H. More than 1,000 cases of total parathyroidectomy with forearm autograft for renal hyperparathyroidism. Am J Kidney Dis. 2001 Oct;38(4 Suppl 1):S168-71. doi: 10.1053/ajkd.2001.27432. PMID 11576947
- [Result] Schneider R, Slater EP, Karakas E, Bartsch DK, Schlosser K. Initial parathyroid surgery in 606 patients with renal hyperparathyroidism. World J Surg. 2012 Feb;36(2):318-26. doi: 10.1007/s00268-011-1392-0. PMID 22202993